CLINICAL TRIAL: NCT06353321
Title: Non-significant Risk (NSR) Study of [68Ga]-PSMA-11 (Illuccix) as a BgRT BioGuide on the RefleXion X1 System in Patients Already Undergoing Diagnostic PET (Positron Emission Tomography) PSMA (Prostate Specific Membrane Antigen) Imaging
Brief Title: Non-significant Risk (NSR) Study of [68Ga]-PSMA-11 (Illuccix) as a BgRT BioGuide on RefleXion X1
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: RefleXion Medical (Industry)
Responsible Party: Principal Investigator, Neil Desai, Principal Investigator, University of Texas Southwestern Medical Center
Other Study IDs: STU-2024-0024
Record Dates: First submitted 2024-03-26; First posted 2024-04-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Single group non blinded: Single Center Study, pilot/feasibility, private for profit observational study
  Interventions: Diagnostic Test: PET-CT imaging subsystem of the RefleXion X1 System Device

INTERVENTIONS:
Diagnostic Test: PET-CT imaging subsystem of the RefleXion X1 System Device — Imaging performed only on the X1 platform immediately following already planned imaging using Illuccix for standard of care indications in men with prostate cancer of various stages, in order to assess performance of the X1 in comparison to diagnostic imaging scanners

SUMMARY:
To qualitatively determine the imaging performance of PET-CT imaging subsystem of the RefleXion X1 System Device in patients undergoing standard-of-care (SOC) [68Ga]-PSMA-11 PET-CT using Illuccix on the same day.

DETAILED DESCRIPTION:
In this non-significant risk (NSR) study, investigators will perform imaging only (no treatment) on the X1 platform immediately following an already planned PET/CT diagnostic imaging using Illuccix for standard of care indications in men with prostate cancer of various stages. This approach will be used to assess imaging performance of the X1 in comparison to diagnostic imaging scanners. Evidence from this study will supplement and enhance technical understanding of the PSMA-11-guided BgRT delivery in the setting of prostate cancer. As such, the patient population selected for this investigation is meant to optimally represent the spectrum of cases, with respect to motion and radiographic environment that a radiation oncologist may encounter in practice.

ELIGIBILITY:
Inclusion Criteria:

* Men with prostate adenocarcinoma undergoing standard of care PSMA-PET imaging for initial staging or re-staging at suspected relapse/progression

Exclusion Criteria:

* 1. Known psychiatric or substance abuse disorder which in the opinion of the investigator would interfere with study conduct

  2. Patient weight exceeding 450 lb (weight limit of RefleXion X1 system)

  3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Males with prostate adenocarcinoma undergoing standard of care PSMA-PET imaging
Study Population: The patient population selected for this investigation is meant to optimally represent the spectrum of cases, with respect to motion and radiographic environment that a radiation oncologist may encounter in practice.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-12-12 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
Qualitative assessment of RefleXion X1 imaging performance with Illuccix PSMA PET imaging agent immediately following a standard of care Illuccix PET/CT | From time of Reflexion scan to 48 hours after scan for adverse event evaluation
  Qualitative imaging performance of the PET subsystem on the X1 system for detect PSMA-11 68Ga (Illuccix)-avid lesions (primary and metastatic) in patients with prostate cancer, relative to diagnostic [68Ga]-PSMA-11 PET-CT.
  This will be assessed by the enrolling investigator with the following question:
  Is there an Illuccix (PSMA-11 Ga68) avid target that correlates to the tumor location on the registered CT image? (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Desai, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Ut Southwestern Medical Center, Dallas, Texas, United States